CLINICAL TRIAL: NCT00542191
Title: Phase II Trial of Neoadjuvant Metronomic Chemotherapy in Triple-Negative Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Enrollment Completed
Sponsor: Leo W. Jenkins Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LJCC 07-03
Record Dates: First submitted 2007-10-09; First posted 2007-10-10 (Estimated); Results first posted 2019-09-10 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Breast Cancer
Keywords: Triple negative (ER/PR negative; HER2 negative)
MeSH Terms: conditions — Breast Neoplasms | interventions — Doxorubicin; Cyclophosphamide; Paclitaxel; Carboplatin; Administration, Metronomic; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Neoadjuvant metronomic AC followed by weekly TC (Experimental): Neoadjuvant chemotherapy with metronomic AC followed by weekly TC then surgery
  Interventions: Drug: Doxorubicin / Cyclophosphamide / Paclitaxel / Carboplatin; Procedure: Definitive Surgery; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Doxorubicin / Cyclophosphamide / Paclitaxel / Carboplatin — DOXORUBICIN 24mg/m2 IV plus CYCLOPHOSPHAMIDE 60mg/m2 PO weekly x 12 successive weeks followed by PACLITAXEL 80mg/m2 IV over 1 hour plus CARBOPLATIN AUC 2 IV weekly x 12 successive weeks
  Other Names: Metronomic
Procedure: Definitive Surgery — Standard of care definitive surgery as determined by medical provider
Radiation: Radiotherapy — Standard of care RADIATION THERAPY as indicated

SUMMARY:
This neoadjuvant chemotherapy protocol focusing on "triple-negative" breast cancers alone will gather a foundation of primary tumor and axillary lymph nodal response to primary chemotherapy and ongoing correlated disease-free (DFS) and overall survival (OS) outcome data. This comparative data can then be used in building subsequent trials.

DETAILED DESCRIPTION:
Women with a diagnosed "triple-negative" proxy of basal-like breast cancer confirmed on a core biopsy and larger than 2 cm will be treated neoadjuvantly with the Livingston metronomic regimen of 12 weeks of weekly doxorubicin 24 mg/m2 and daily oral cyclophosphamide 60 mg/m2 followed by 12 successive weeks of taxol 80 mg/m2 and carboplatin AUC 2. Although clinical response will be evaluated prior to surgery, the primary end-point is the pathologic response. Secondary end-points will be DFS and OS based upon standard of care surveillance. A pathologic complete response (pCR) will require no histologic evidence of residual malignant cells seen in the primary tumor area specimen or the lymph nodes. Standard of care surgery and radiation therapy will be undertaken.

ELIGIBILITY:
Inclusion Criteria:

* Women with Estrogen Receptor (ER), Progesterone Receptor (PR),and HER2 negative invasive breast cancer confirmed on core biopsy.(Note: HER2 negative by FISH preferred; HER2 0 or 1+ by IHC acceptable)
* Primary tumor size 2cm or greater by physical exam or radiographic measurements.(Note: Locally advanced T4 or inflammatory breast cancer is eligible.)
* Assessment of pre-treatment axillary lymph nodal status (Note: FNA biopsy if palpable or sentinel lymph node biopsy (SLNB) if not palpable preferred; clinical exam acceptable.)
* Absolute neutrophil count > 1500 mm3 and platelet count > 100,000 mm3
* Normal myocardial left ventricular function
* Serum creatinine < 2.0 mg/dl
* Total bilirubin and AST < 3X upper limits normal

Exclusion Criteria:

* Recurrent or metastatic breast cancer findings (Note: If oncologically felt to be a second breast primary, patient eligible for this protocol)
* Another active cancer present
* Medical contraindications to chemotherapy or surgery
* First trimester pregnancy
* Breast feeding

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-07; Primary Completion 2016-08-02 (Actual); Study Completion 2016-08-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Walker, MD, Principal Investigator — Brody School of Medicine at East Carolina University
Locations (1):
- Brody School of Medicine at East Carolina University, Greenville, North Carolina, United States

REFERENCES:
- [Background] Sorlie T, Perou CM, Tibshirani R, Aas T, Geisler S, Johnsen H, Hastie T, Eisen MB, van de Rijn M, Jeffrey SS, Thorsen T, Quist H, Matese JC, Brown PO, Botstein D, Lonning PE, Borresen-Dale AL. Gene expression patterns of breast carcinomas distinguish tumor subclasses with clinical implications. Proc Natl Acad Sci U S A. 2001 Sep 11;98(19):10869-74. doi: 10.1073/pnas.191367098. PMID 11553815
- [Background] Perou CM, Sorlie T, Eisen MB, van de Rijn M, Jeffrey SS, Rees CA, Pollack JR, Ross DT, Johnsen H, Akslen LA, Fluge O, Pergamenschikov A, Williams C, Zhu SX, Lonning PE, Borresen-Dale AL, Brown PO, Botstein D. Molecular portraits of human breast tumours. Nature. 2000 Aug 17;406(6797):747-52. doi: 10.1038/35021093. PMID 10963602
- [Background] Sotiriou C, Neo SY, McShane LM, Korn EL, Long PM, Jazaeri A, Martiat P, Fox SB, Harris AL, Liu ET. Breast cancer classification and prognosis based on gene expression profiles from a population-based study. Proc Natl Acad Sci U S A. 2003 Sep 2;100(18):10393-8. doi: 10.1073/pnas.1732912100. Epub 2003 Aug 13. PMID 12917485
- [Background] Brenton JD, Carey LA, Ahmed AA, Caldas C. Molecular classification and molecular forecasting of breast cancer: ready for clinical application? J Clin Oncol. 2005 Oct 10;23(29):7350-60. doi: 10.1200/JCO.2005.03.3845. Epub 2005 Sep 6. PMID 16145060
- [Background] Nielsen TO, Hsu FD, Jensen K, Cheang M, Karaca G, Hu Z, Hernandez-Boussard T, Livasy C, Cowan D, Dressler L, Akslen LA, Ragaz J, Gown AM, Gilks CB, van de Rijn M, Perou CM. Immunohistochemical and clinical characterization of the basal-like subtype of invasive breast carcinoma. Clin Cancer Res. 2004 Aug 15;10(16):5367-74. doi: 10.1158/1078-0432.CCR-04-0220. PMID 15328174
- [Background] Chang HY, Nuyten DS, Sneddon JB, Hastie T, Tibshirani R, Sorlie T, Dai H, He YD, van't Veer LJ, Bartelink H, van de Rijn M, Brown PO, van de Vijver MJ. Robustness, scalability, and integration of a wound-response gene expression signature in predicting breast cancer survival. Proc Natl Acad Sci U S A. 2005 Mar 8;102(10):3738-43. doi: 10.1073/pnas.0409462102. Epub 2005 Feb 8. PMID 15701700
- [Background] Turner N, Tutt A, Ashworth A. Hallmarks of 'BRCAness' in sporadic cancers. Nat Rev Cancer. 2004 Oct;4(10):814-9. doi: 10.1038/nrc1457. PMID 15510162
- [Background] Carey LA, Perou CM, Livasy CA, Dressler LG, Cowan D, Conway K, Karaca G, Troester MA, Tse CK, Edmiston S, Deming SL, Geradts J, Cheang MC, Nielsen TO, Moorman PG, Earp HS, Millikan RC. Race, breast cancer subtypes, and survival in the Carolina Breast Cancer Study. JAMA. 2006 Jun 7;295(21):2492-502. doi: 10.1001/jama.295.21.2492. PMID 16757721
- [Background] Berry DA, Cirrincione C, Henderson IC, Citron ML, Budman DR, Goldstein LJ, Martino S, Perez EA, Muss HB, Norton L, Hudis C, Winer EP. Estrogen-receptor status and outcomes of modern chemotherapy for patients with node-positive breast cancer. JAMA. 2006 Apr 12;295(14):1658-67. doi: 10.1001/jama.295.14.1658. PMID 16609087
- [Background] Kennedy RD, Quinn JE, Mullan PB, Johnston PG, Harkin DP. The role of BRCA1 in the cellular response to chemotherapy. J Natl Cancer Inst. 2004 Nov 17;96(22):1659-68. doi: 10.1093/jnci/djh312. PMID 15547178
- [Background] Kerbel RS, Klement G, Pritchard KI, Kamen B. Continuous low-dose anti-angiogenic/ metronomic chemotherapy: from the research laboratory into the oncology clinic. Ann Oncol. 2002 Jan;13(1):12-5. doi: 10.1093/annonc/mdf093. No abstract available. PMID 11863092
- [Background] Robert N, Leyland-Jones B, Asmar L, Belt R, Ilegbodu D, Loesch D, Raju R, Valentine E, Sayre R, Cobleigh M, Albain K, McCullough C, Fuchs L, Slamon D. Randomized phase III study of trastuzumab, paclitaxel, and carboplatin compared with trastuzumab and paclitaxel in women with HER-2-overexpressing metastatic breast cancer. J Clin Oncol. 2006 Jun 20;24(18):2786-92. doi: 10.1200/JCO.2005.04.1764. PMID 16782917
- [Background] Perez EA, Suman VJ, Rowland KM, Ingle JN, Salim M, Loprinzi CL, Flynn PJ, Mailliard JA, Kardinal CG, Krook JE, Thrower AR, Visscher DW, Jenkins RB. Two concurrent phase II trials of paclitaxel/carboplatin/trastuzumab (weekly or every-3-week schedule) as first-line therapy in women with HER2-overexpressing metastatic breast cancer: NCCTG study 983252. Clin Breast Cancer. 2005 Dec;6(5):425-32. doi: 10.3816/CBC.2005.n.047. PMID 16381626
- [Background] Kaufmann M, Hortobagyi GN, Goldhirsch A, Scholl S, Makris A, Valagussa P, Blohmer JU, Eiermann W, Jackesz R, Jonat W, Lebeau A, Loibl S, Miller W, Seeber S, Semiglazov V, Smith R, Souchon R, Stearns V, Untch M, von Minckwitz G. Recommendations from an international expert panel on the use of neoadjuvant (primary) systemic treatment of operable breast cancer: an update. J Clin Oncol. 2006 Apr 20;24(12):1940-9. doi: 10.1200/JCO.2005.02.6187. PMID 16622270
- [Background] Hennessy BT, Hortobagyi GN, Rouzier R, Kuerer H, Sneige N, Buzdar AU, Kau SW, Fornage B, Sahin A, Broglio K, Singletary SE, Valero V. Outcome after pathologic complete eradication of cytologically proven breast cancer axillary node metastases following primary chemotherapy. J Clin Oncol. 2005 Dec 20;23(36):9304-11. doi: 10.1200/JCO.2005.02.5023. PMID 16361629
- [Background] Buzdar AU, Ibrahim NK, Francis D, Booser DJ, Thomas ES, Theriault RL, Pusztai L, Green MC, Arun BK, Giordano SH, Cristofanilli M, Frye DK, Smith TL, Hunt KK, Singletary SE, Sahin AA, Ewer MS, Buchholz TA, Berry D, Hortobagyi GN. Significantly higher pathologic complete remission rate after neoadjuvant therapy with trastuzumab, paclitaxel, and epirubicin chemotherapy: results of a randomized trial in human epidermal growth factor receptor 2-positive operable breast cancer. J Clin Oncol. 2005 Jun 1;23(16):3676-85. doi: 10.1200/JCO.2005.07.032. Epub 2005 Feb 28. PMID 15738535
- [Background] Rouzier R, Anderson K, Hess KR, et al: Basal and luminal types of breast cancer defined by gene expression patterns respond differently to neoadjuvant chemotherapy. San Antonio Breast Cancer Symposium. San Antonio, TX, 2004 (abstr 1023)
- [Background] Carey LA, Dees EC, Sawyer L, et al: The triple negative paradox: Primary tumor chemosensitivity of the basal-like breast cancer (BBC) phenotype. San Antonio Breast Cancer Symposium. San Antonio, TX, 2004 (abstr 1023)
- [Background] Jacquemier J, Penault-Llorca F, Mnif H, et al: Identification of a basal-like subtype and comparative effect of epirubicin-based chemotherapy and sequential epirubicin followed by docetaxel chemotherapy in the PACS 01 breast cancer trial: 33 markers studied on tissue microarrays (TMA). J Clin Oncol 2006 (suppl; abstr 509)
- [Background] Hudis C, Citron M, Berry D, et al: Five-year follow-up of INT C9741: dose-dense chemotherapy is safe and effective. San Antonio Breast Cancer Symposium. San Antonio, TX, 2005 (abstr 41)
- [Background] Ellis GK, Livingston RB, Rinn K, et al: Pilot adjuvant study: 12 weeks of dose dense doxorubicin with scheduled G-CSF support followed by 4 cycles of docetaxel. J Clin Oncol 2003 (suppl; abstr 148)
- [Background] Ellis GK, Barlow WE, Gralow JR, Hortobagyi GN, Russell CA, Royce ME, Perez EA, Lew D, Livingston RB. Phase III comparison of standard doxorubicin and cyclophosphamide versus weekly doxorubicin and daily oral cyclophosphamide plus granulocyte colony-stimulating factor as neoadjuvant therapy for inflammatory and locally advanced breast cancer: SWOG 0012. J Clin Oncol. 2011 Mar 10;29(8):1014-21. doi: 10.1200/JCO.2009.27.6543. Epub 2011 Jan 10. PMID 21220618

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase II Trial Neoadjuvant Metronomic AC Followed by TC: Doxorubicin / Cyclophosphamide / Paclitaxel / Carboplatin: DOXORUBICIN 24mg/m2 IV plus CYCLOPHOSPHAMIDE 60mg/m2 PO weekly x 12 successive weeks followed by PACLITAXEL 80mg/m2 IV over 1 hour plus CARBOPLATIN AUC 2 IV weekly x 12 successive weeks
  Definitive Surgery: Standard of care definitive surgery as determined by medical provider
  Radiotherapy: Standard of care RADIATION THERAPY as indicated
Period: Overall Study
Arm/Group | Phase II Trial Neoadjuvant Metronomic AC Followed by TC
Started | 21
Completed | 18
Not Completed | 3
Not completed — Death | 3

BASELINE CHARACTERISTICS:
Population: Slow accrual
Groups:
- Single Arm Study; Taxol, XRT, Gemzar and Carbo: Doxorubicin / Cyclophosphamide / Paclitaxel / Carboplatin: DOXORUBICIN 24mg/m2 IV plus CYCLOPHOSPHAMIDE 60mg/m2 PO weekly x 12 successive weeks followed by PACLITAXEL 80mg/m2 IV over 1 hour plus CARBOPLATIN AUC 2 IV weekly x 12 successive weeks
  Definitive Surgery: Standard of care definitive surgery as determined by medical provider
  Radiotherapy: Standard of care RADIATION THERAPY as indicated
Arm/Group | Single Arm Study; Taxol, XRT, Gemzar and Carbo
Number analyzed (Participants) | 21
Age, Continuous [Median (Full Range); unit: years] | 50 [32 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: 1) Pathologic Response
Description: Pathologic measurement post-surgery viable primary tumor mass
Time Frame: Upon completion therapy after surgery
Population: Study closed to accrual - not enough participants to participate.
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm Study; Taxol, XRT, Gemzar and Carbo
Number analyzed (Participants) | 18
Participants | 15

ADVERSE EVENTS:
Time Frame: Upon completion neoadjuvant chemotherapy and surgery
Arm/Group | Single Arm Study; Taxol, XRT, Gemzar and Carbo
All-Cause Mortality (participants affected / at risk) | 3/21
Serious Adverse Events (participants affected / at risk) | 3/21
Other Adverse Events (participants affected / at risk) | 0/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm Study; Taxol, XRT, Gemzar and Carbo (N=21)
sepsis (Infections and infestations) | 2 (2)
pulmonary embolus (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes